CLINICAL TRIAL: NCT02969629
Title: The Effects of the Dopamine Agonist (Apomorphine) on Experimental and Clinical Pain in Patients With Chronic Radicular Pain: a Randomized, Double-blind, Placebo-controlled, Cross-over Study
Brief Title: The Effects of Apomorphine on Experimental and Clinical Pain in Patients With Chronic Radicular Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Eisenberg Elon MD, Head of pain research unit, Institute of pain, Rambam Health Care Campus
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0234-11-RMB
Record Dates: First submitted 2016-09-14; First posted 2016-11-21 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Apomorphine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- apomorphine (Experimental): 1.5 mg apomorphine, administered subcutaneously
  Interventions: Drug: Apomorphine
- Normal saline (Placebo Comparator): saline, administered subcutaneously
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Apomorphine
  Arms: apomorphine
Drug: Normal Saline
  Arms: Normal saline

SUMMARY:
The study aimed to explore the effect of the dopamine agonist apomorphine on spontaneous pain intensity and evoked cold clinical and experimental pain in patients with lumbar radicular neuropathic pain (NP). Patients received either apomorphine or placebo in a randomized double-blinded manner.

DETAILED DESCRIPTION:
Although evidence suggests that dopaminergic systems are involved in pain processing, the efficacy of dopaminergic interventions in reducing pain remains questionable. This randomized, double blinded, placebo-controlled, cross-over study was aimed to explore the effect of the dopamine agonist apomorphine on spontaneous pain intensity and evoked cold clinical and experimental pain in patients with lumbar radicular neuropathic pain (NP).

Data was collected from 35 patients (18 men, mean age 56.2±13.1 years). The following five pain measures were tested before (baseline) and 30, 75 and 120 min subsequent to subcutaneous injection of 1.5 mg apomorphine or placebo in two separate sessions: spontaneous pain intensity, threshold and tolerance to cold pain in the most painful site in the affected leg and in a remote healthy site in the dominant hand.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of radicular pain for at least 3 months;
2. Average pain level during the last week prior to enrollment > 40 (0-100);
3. No use of a new analgesic drug within 30 days prior to entry to the study and
4. Adults who were capable of understanding the purpose and instructions of the study and signing an informed consent.

Exclusion Criteria:

1. Pregnancy or breastfeeding;
2. Presence of Parkinson's disease or any other extra-pyramidal diseases;
3. History of allergy to the investigational drugs: Apomorphine or Domperidone;
4. History of polyneuropathy and
5. Respiratory depression, dementia, psychotic diseases or hepatic insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Experimental and clinical cold pain tolerance measured in seconds | Up to 120 minutes after drug administration

SECONDARY OUTCOMES:
Experimental and clinical cold pain threshold measured in seconds | Up to 120 minutes after drug administration
Spontaneous clinical pain intensity measured on a numeric pain scale (NPS, 0-100) | Up to 120 minutes after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Elon Eisenberg, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.